CLINICAL TRIAL: NCT00088621
Title: An Open-Label, Multicenter, Twelve-Month Study of Safety and Tolerability in the Treatment of Schizophrenia
Brief Title: A Study to Test the Safety and Tolerability of a New Medication in the Treatment of Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1050199
Record Dates: First submitted 2004-07-30; First posted 2004-08-02 (Estimated); Results first posted 2011-05-06 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-03

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Latuda; Lurasidone
MeSH Terms: conditions — Schizophrenia | interventions — Lurasidone Hydrochloride; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lurasidone 80 mg tablet (Experimental): Lurasidone 80mg oral tablet taken once a day
  Interventions: Drug: Lurasidone 80mg tablet

INTERVENTIONS:
Drug: Lurasidone 80mg tablet
  Other Names: Lurasidone

SUMMARY:
A 1-year outpatient study to test the safety and tolerability of a new medication in the treatment of schizophrenia

DETAILED DESCRIPTION:
Study will evaluate long-term safety and tolerability of a new compound in the treatment of patients with schizophrenia as assessed by adverse events (AEs), measures of extra pyramidal symptoms (EPS; Abnormal Involuntary Movement Scale [AIMS], Barnes Akathisia Scale [BAS], and Simpson-Angus Rating Scale [SAS]), vital sign measurements, electrocardiograms (ECGs), clinical laboratory evaluations.

ELIGIBILITY:
* Patients must have participated in study D1050196 (A Study to Test the Effectiveness and Safety of a New Medication in the Treatment of Schizophrenia) and either:
* Successfully completed
* OR
* Patients must have been discontinued after a minimum of 2 weeks of treatment due to lack of efficacy

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2004-07; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Sumitomo Pharma America, Inc.
Locations (21):
- United States (21):
  - Birmingham Psychiatry Pharmaceutical, Birmingham, Alabama
  - Summit Research Group, Little Rock, Arkansas
  - Comprehensive NeuroScience, Cerritos, California
  - Collaborative Neuro Science Network, Inc., Garden Grove, California
  - Optimum Health Services, La Mesa, California
  - California Clinical Trials, San Diego, California
  - CA Neutopsychopharmacology Clinical Research Institute (CNRI), San Diego, California
  - Pacific Clinical Research, Upland, California
  - Comprehensive NeuroScience, Inc, Washington D.C., District of Columbia
  - Segal Institute for Clinical Research, Fort Lauderdale, Florida
  - Segal Institute for Clinical Research, North Miami, Florida
  - University of South Florida, Department of Psychiatry and Behavioral Medicine, Tampa, Florida
  - Comprehensive Neuroscience, Inc., Hoffman Estates, Illinois
  - Las Vegas, Nevada
  - CNS Research Institute, Clementon, New Jersey
  - Quantum Clinical Services Group, Philadelphia, Pennsylvania
  - Community Clinical Research, Austin, Texas
  - Future Search Trials, Austin, Texas
  - Claghorn Lesem Research Clinic, Inc., Bellaire, Texas
  - InSite Clinical Research, DeSoto, Texas
  - CBH Health, L.L.C - Dominion Hospital, Falls Church, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Lurasidone 80 mg: Lurasidone 80mg oral tablet. The number of subjects that represent the participant flow is based on the number of subjects that entered the extension study which is 61 subjects.
Period: Overall Study
Arm/Group | Lurasidone 80 mg
Started | 61
Completed | 7
Not Completed | 54

BASELINE CHARACTERISTICS:
Groups:
- Lurasidone 80 mg: Lurasidone 80mg oral tablet. The number of subjects that represent the baseline must have taken 1 dose of study medication and had post-baseline assessment. 2 subjects were randomized and did not take study medication and thus 59 subjects is listed in the baseline group.
Arm/Group | Lurasidone 80 mg
Number analyzed (Participants) | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.3 (11.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 44
Region of Enrollment [Number; unit: participants]
  United States | 59

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With an Adverse Events in a One Year Open Label Lurasidone Study
Time Frame: 1 year
Population: Number of subjects that entered into the extension trial.
Measure: Number; unit: participants
Arm/Group | Lurasidone 80 mg
Number analyzed (Participants) | 61
participants | 59

ADVERSE EVENTS:
Arm/Group | Lurasidone 80 mg
Serious Adverse Events (participants affected / at risk) | 12/59
Other Adverse Events (participants affected / at risk) | 18/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lurasidone 80 mg (N=59)
Pericardial Effusion (Cardiac disorders) | 1 (1)
Orchitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 1 (1)
Schizophrenia (Psychiatric disorders) | 8 (8)
Self Injurious Behavior (Psychiatric disorders) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1)
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lurasidone 80 mg (N=59)
Nausea (Gastrointestinal disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 3 (3)
Bronchitis (Infections and infestations) | 4 (4)
Nasopharyngitis (Infections and infestations) | 3 (3)
Upper Respiratory Tract Infection (Infections and infestations) | 3 (3)
Weight Decreased (Investigations) | 3 (3)
Weight Increased (Investigations) | 4 (4)
Sedation (Nervous system disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No